CLINICAL TRIAL: NCT03788161
Title: Effects of Virtual Reality on Post-Needling Soreness After Dry Needling of Trigger Points in the Extensor Carpi Radialis Brevis
Brief Title: Virtual Reality and Post-dry Needling Soreness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, César Fernández-de-las-Peñas, Director of Department, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: URJC1509201810418
Record Dates: First submitted 2018-12-22; First posted 2018-12-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Healthy; Epicondylitis of the Elbow
Keywords: trigger points; virtual reality; Dry needling

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real Virtual Reality (Experimental): Participants will receive a distraction by playing a game of virtual reality with a 3D application
  Interventions: Other: Real Virtual Reality
- Placebo Virtual Reality (Placebo Comparator): Participants will receive a placebo distraction with a game of virtual reality with a 3D application without functioning
  Interventions: Other: Placebo Virtual Reality

INTERVENTIONS:
Other: Real Virtual Reality — Participants will receive a distraction by playing a game of virtual reality with a 3D application
  Arms: Real Virtual Reality
Other: Placebo Virtual Reality — Participants will receive a placebo distraction with a game of virtual reality with a 3D application without functioning
  Arms: Placebo Virtual Reality

SUMMARY:
Application of trigger point dry needling can induce post-dry needling soreness. This is not a negative experience, but sometimes some patients want to reduce it as much as possible. Different therapeutic strategies targeting to decrease post-dry needling soreness need to be investigated. Previous studies have investigated spray and stretch, ischemic compression or low-load eccentric exercise as post-needling intervention procedures. There is increasing evidence supporting the role of descending pain inhibition mechanisms for paon control. The application of virtual reality as a distraction technique could active brain mechanisms during dry needling. Therefore, the objective of this study will be to investigate the effects of playing virtual reality during the application of dry needling on post-needling soreness over trigger points in the extensor carpi radialis brevis muscle. A secondary aim will be to determine the prognostic role of baseline scores of pressure pain sensitivity, related-disability, anxiety and catastrophizing levels.

ELIGIBILITY:
Inclusion Criteria for pain-free participants:

* no history of upper quadrant pain symptoms the year preceding the study
* no history of upper quadrant surgery
* presence of a latent trigger point in the extensor carpi radialis brevis muscle

Inclusion criteria for patients with elbow pain:

* pain over the lateral side of the elbow;
* pain on palpation over the lateral epicondyle or the associated common wrist extensor tendon;
* elbow pain with either resisted static contraction or stretching of the wrist extensor muscles.
* presence of an active trigger point in the extensor carpi radialis brevis muscle

Exclusion Criteria:

* bilateral symptoms;
* older than 50 years of age;
* previous surgery or steroid injections;
* other diagnoses of upper extremity (shoulder pathology, cervical radiculopathy, cervical whiplash);
* history of cervical or upper extremity trauma;
* history of musculoskeletal medical conditions (rheumatoid arthritis, fibromyalgia);

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Changes in post-dry needling pain assessed with a numerical pain rate scale before and after the intervention | Baseline, 5 minutes after, 12 hours after, 24 hours after, 36 hours after, 48 hours after, and 72 hours after treatment
  A numerical Pain Rate Scale (NPRS, 0-10) will be used to record post-dry needling soreness and pain

SECONDARY OUTCOMES:
Baseline score of upper extremity related-disability assessed with the Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire | Baseline
  The DASH questionaire consists of 30-items assessing: 1, degree of difficulty during the preceding week in performing physical activities because of problems in the upper extremity (21 items); 2, severity of each pain symptom, activity-related pain, tingling, weakness, and stiffness (5 items); and, 3, the problem's effect on social activities, work, and sleep, and its psychological impact (4 items). Each item is answered on a 5-points scale ranging from 1 (no difficulty to perform, no symptom, or no impact) to 5 (unable to do, very severe symptom, or high impact). Responses are summed to form a raw score that is converted to a 0 to 100 scale where higher scores reflect greater related-disability.
Baseline data on pressure pain sensitivity assessed with a pressure algometer | Baseline
  Pressure pain thresholds over the cervical spine, the lateral epicondyle and the tibialis anterior muscle will be assessed with a pressure algometer at baseline
Baseline anxiety levels as assessed with the State-Trait Anxiety Inventory (STAI) questionnaire | Baseline
  The STAI is a 40 items scale assessing separate dimensions of state anxiety (items l-20, STAI-S) and trait anxiety (items 21-40, STAI-T). The STAI-S items assess relatively enduring symptoms of anxiety. Participants use a 4-points response scale ranging from "not at all" to "very much", to indicate the extent to which they experience each emotion. The STAI-T scale measures a stable propensity to experience anxiety, and tendencies to perceive stressful situations as threatening. It consists of 20 statements requiring individuals to rate how they generally feel on a 4-points scale. In both scales, higher scores indicate greater state or trait anxiety.
Catastrophizing belief as assessed with the Pain Catastrophizing Scale | Baseline
  The Pain Catastrophizing Scale will be used for determining baseline participant's propensity to catastrophize about pain. It consists of 13-items evaluating the three components of catastrophizing: rumination, magnification and helplessness.

CONTACTS AND LOCATIONS:
Locations (1):
- Cesar Fernandez-de-Las-Peñas, Alcorcón, Madrid, Spain